CLINICAL TRIAL: NCT04587076
Title: Evaluation of Protein Intake, Vitamin, Mineral, and Trace Element Supplementation After Bariatric Surgery According to the German S3 Guidelines - What Effects do Age, Sex, and Socio-economic Status Have on Adherence?
Brief Title: Evaluation of Protein Intake and Micronutrient Supplementation After Bariatric Surgery
Acronym: BOP
Status: Completed | Type: Observational
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Other Study IDs: BB 080/19
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Protein Malnutrition; Vitamin Deficiency; Mineral Deficiency; Trace Element Deficiency; Obesity; Obesity, Morbid
Keywords: Gastric Bypass; Gastric Sleeve
MeSH Terms: conditions — Kwashiorkor; Avitaminosis; Obesity; Obesity, Morbid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Faeces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obesity is a chronic disease in which accumulation of excess body fat can result in impaired health. In cases of severe obesity, weight loss surgery can be necessary as a treatment. There are different forms of surgery but the common basic principle is to restrict food intake and decrease the absorption of food in the stomach and intestines. As a consequence, there is a higher risk of developing nutrient deficiency after surgery and supplementation of protein, vitamins, and minerals can be necessary. This study evaluates intakes of protein, vitamins, and minerals in patients with weight loss surgery and compares them to recommended intakes. Further, this study looks at the role of age, sex, and socioeconomic status in this context.

DETAILED DESCRIPTION:
Obesity is defined by the World Health Organization as abnormal or excessive fat accumulation that may impair health. These days, bariatric surgery is considered the most effective treatment of morbid obesity. In the last decade, the number of bariatric surgeries performed worldwide constantly increased. Common bariatric surgery procedures include gastric bypass, sleeve gastrectomy, adjustable gastric band, and biliopancreatic diversion with duodenal switch. After surgery, weight loss is induced by a reduced food volume the stomach can hold, malabsorption of nutrients, or by a combination of both mechanisms. In consequence, patients with bariatric surgery have an increased risk of developing nutrient deficiency. Therefore, guidelines recommend supplementation of critical nutrients, i.e. protein, vitamins, and minerals, after bariatric surgery. This study assesses intake of these nutrients in patients with bariatric surgery based on the recommendations provided by the German S3 Guideline Group on the Surgical Treatment of Obesity and Metabolic Diseases. In particular, this study assesses the association of therapy adherence with age, sex, and socioeconomic status.

ELIGIBILITY:
Inclusion Criteria:

* Sleeve gastrectomy (postoperative)
* Roux-en-Y gastric Bypass (postoperative)
* Postoperative period > 6 month

Exclusion Criteria:

* Missing consent
* Pregnancy
* Malignant tumor
* Implanted pacemaker
* Any other serious primary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were recruited at University Medicine Greifswald, a medical center with expertise in obesity Treatment located in Northeast Germany. Patients meeting the study's eligibilty criteria who attended their routine postoperative care visits after bariatric surgery were approached for study participation.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Therapy Adherence Across Groups of Socio-Economic Status | Baseline
  Number of recommendations followed by the patients according to the recommendations provided by the German S3 Guidelines across groups of socio-economic status.

SECONDARY OUTCOMES:
Therapy Adherence Across Age Groups | Baseline
  Number of recommendations followed by the patients according to the recommendations provided by the German S3 Guidelines across age groups.
Therapy Adherence Across Sexes | Baseline
  Number of recommendations followed by the patients according to the recommendations provided by the German S3 Guidelines across sexes.
Improvement of Deficiency Symptoms | Baseline
  Determination of improvement of deficiency symptoms through adequate supplementation after bariatric surgery
Body Weight | Baseline
  Determination of body weight measured in kilograms
Body Height | Baseline
  Determination of body height measured in centimeters
Body Mass Index | Baseline
  Determination of body mass index measured in kg/m^2 (calculated from the values obtained for body weight and height)
Waist Circumference | Baseline
  Determination of waist circumference measured in centimeters
Hip Circumference | Baseline
  Determination of hip circumference measured in centimeters
Waist-to-Hip Ratio | Baseline
  Determination of waist-to-hip ratio (calculated from the values obtained for waist and hip circumference)
Triceps Skinfold Thickness | Baseline
  Determination of triceps skinfold thickness measured in millimeters
Upper Arm Circumference | Baseline
  Determination of upper arm circumference measured in centimeters
Fat Free Mass | Baseline
  Determination of fat free mass measured by Bioelectrical Impedance Analysis (BIA)
Skeletal Muscle Mass | Baseline
  Determination of skeletal muscle mass measured by Bioelectrical Impedance Analysis (BIA)
Fat Mass | Baseline
  Determination of fat mass measured by Bioelectrical Impedance Analysis (BIA)
Total Body Water | Baseline
  Determination of total body water measured by Bioelectrical Impedance Analysis (BIA)
Extracellular Water | Baseline
  Determination of extracellular water measured by Bioelectrical Impedance Analysis (BIA)
Phase Angle | Baseline
  Determination of phase angle measured by Bioelectrical Impedance Analysis (BIA)
Muscle Strength | Baseline
  Determination of muscle strength assessed by handgrip dynamometry
Systolic Blood Pressure | Baseline
  Determination of systolic blood pressure in mmHg
Diastolic Blood Pressure | Baseline
  Determination of diastolic blood pressure in mmHg
Physical Activity | Baseline
  Determination of metabolic equivalents of task per day and activity level assessed by employment of the German version of the International Physical Activity Questionnaire (IPAQ) Short Form
Energy Intake | Baseline
  Determination of energy intake (kcal/d) assessed by 7-day dietary record
Protein Intake | Baseline
  Determination of protein intake assessed by 7-day dietary record
Fat Intake | Baseline
  Determination of fat intake assessed by 7-day dietary record
Omega-3 Fatty Acid Intake | Baseline
  Determination of omega-3 fatty acid intake assessed by 7-day dietary record
Omega-6 Fatty Acid Intake | Baseline
  Determination of omega-6 fatty acid intake assessed by 7-day dietary record
Carbohydrate Intake | Baseline
  Determination of carbohydrate intake assessed by 7-day dietary record
Dietary Fiber Intake | Baseline
  Determination of dietary fiber intake assessed by 7-day dietary record
Sucrose Intake | Baseline
  Determination of sucrose intake intake assessed by 7-day dietary record
Alcohol Intake | Baseline
  Determination of alcohol intake intake assessed by 7-day dietary record
Diet Quality | Baseline
  Determination of diety quality assessed by 7-day dietary record based on the Alternate Healthy Eating Index 2010 (AHEI-2010) score. Scores range from 0 to 110, with higher scores indicating higher diet quality
Quality of Life Assessment | Baseline
  Quality of life was assessed by employment of the German Short Form-12 Questionnaire, with higher scores indicating better quality of life.
Intestinal Microbiome | Baseline
  Determination of intestinal microbiome composition in comparison to healthy control subjects

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. med. Markus M. Lerch, Principal Investigator — University Medicine Greifswald
Locations (1):
- University Medicine Greifswald, Greifswald, Germany